CLINICAL TRIAL: NCT00799110
Title: Vaccination of Patients With Ovarian Cancer With Dendritic Cell/Tumor Fusions With GM-CSF and Imiquimod
Brief Title: Vaccination of Patients With Ovarian Cancer With Dendritic Cell/Tumor Fusions With Granulocyte Macrophage Colony-stimulating Factor (GM-CSF) and Imiquimod
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Avigan, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-380
Record Dates: First submitted 2008-11-26; First posted 2008-11-27 (Estimated); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cancer; Fallopian Tube Cancer
Keywords: dendritic cells; fusion vaccines; GM-CSF; imiquimod
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 2 (Experimental): Vaccine, GM-CSF and imiquimod,
  Interventions: Drug: GM-CSF; Biological: Dendritic Cell/Tumor Fusion Vaccine; Drug: imiquimod
- Group 1 (Experimental): Vaccination plus GM-CSF
  Interventions: Drug: GM-CSF; Biological: Dendritic Cell/Tumor Fusion Vaccine

INTERVENTIONS:
Drug: GM-CSF — Injections given subcutaneously at the sight of vaccination on the day of the vaccination and for three days afterwards
Biological: Dendritic Cell/Tumor Fusion Vaccine — Given subcutaneously once every three weeks for a total of three vaccines
  Other Names: DC/tumor fusion vaccine
Drug: imiquimod — Cream applied to the skin at the injection sight 2 hours before injection and for 3 days following the injection
  Arms: Group 2

SUMMARY:
This research study is evaluating the effect (good and bad) of a dendritic cell/tumor fusion vaccine in combination with the laboratory made agents GM-CSF and imiquimod on the participants immune system. Another purpose of this study is to determine the type and severity of any side effects associated with this new study vaccine. We will also be evaluating what effect the vaccine has on the participants cancer. Dendritic cell vaccines have already been tested in clinical trials involving participants with many different types of cancer. Dendritic cells are powerful immune-stimulating cells that are normally found in small amounts in the body and are responsible for immune responses against "foreign" substances that enter the body.

DETAILED DESCRIPTION:
* Patients must have undergone therapeutic debulking surgery for independent clinical indications and have tissue frozen and stored under sterile conditions as part of protocol 07-319 (Study of Primary Tumor Harvest for the Purpose of Possible Use in a Future Clinical Trial in Patients with Ovarian, Fallopian Tube, or Primary Peritoneal Cancer)
* Participants will be assigned to one of two study groups. Both groups will undergo a procedure known as leukapheresis by which the white blood cells are removed from the participants blood in order to obtain the dendritic cells. Prior to this procedure participants may receive 4 injections of GM-CSF, which helps increase the white blood cell count.
* If enough cells are obtained during the leukapheresis, tumor cells and dendritic cells will then be fused (mixed) together in the laboratory and divided into the appropriate doses for administration.
* Participants assigned to Group 1 will undergo subcutaneous vaccination with the dendritic cell tumor fusion vaccine. On the day of the vaccine and three days afterwards, they will receive GM-CSF injections at the site of the vaccination. Participants will receive a dose of the vaccine every 3 weeks for a total of 3 vaccinations.
* Participants assigned to Group 2 will undergo subcutaneous vaccination with the dendritic cell tumor fusion vaccine. On the day of the vaccine and three days afterwards, they will receive GM-CSF injection at the site of the vaccination. Additionally, imiquimod cream will be applied to the skin at the injection sight 2 hours before the vaccine administration. Participants will continue to apply imiquimod cream at the site of vaccination for 3 days following the injection. Participants will receive a dose of the vaccine every 3 weeks for a total of 3 vaccinations.

ELIGIBILITY:
Inclusion criteria at time of initial enrollment:

* Patients must have undergone therapeutic debulking surgery for independent clinical indications and have tissue frozen and stored under sterile conditions as part of protocol 07-319 (Study of Primary Tumor Harvest for the Purpose of Possible Use in a Future Clinical Trial in Patients with Ovarian, Fallopian Tube, or Primary Peritoneal Cancer)
* Patients with histologically proven stage III or IV ovarian, fallopian tube or primary peritoneal serous carcinoma (or patients of any stage with recurrent disease) who demonstrate lack of disease progression as determined by clinical assessment as well as CA-125 levels and/or radiographic assessment
* Patients must have ECOG performance status of 0-2 with greater than six week life expectancy.
* All patients must be informed of the investigational nature of this study and must give written informed consent in accordance with institutional and federal guidelines.
* Laboratories:WBC > 2.0 X 103/uL, Platelets > 50,000/uL, Bilirubin < 2.0 mg/dL, Creatinine <2.0 mg/dL, AST/ALT < 2.5 x ULN

Eligibility criteria prior to first vaccination

At a maximum of twelve weeks after the last dose of chemotherapy, patients must fulfill the following criteria:

* Complete clinical response after first-line chemotherapy for newly-diagnosed patients, or after second-line chemotherapy for relapsed patients who require secondary cytoreduction.**
* Asymptomatic, low volume disease not requiring further chemotherapy prior to initiating vaccination

  ** Complete clinical response is defined as normal exam, normal CT scan, and normal CA-125 level. Tumor tissue for relapsed patients would be obtained under informed consent at the time of a secondary surgical debulking, which would be performed as part of standard relapse management in appropriate patients.
* Resolution of all chemotherapy related grade III-IV toxicity
* Laboratories:WBC > 2.0 X 103/uL, Platelets > 50,000/uL, Bilirubin < 2.0 mg/dL Creatinine <2.0 mg/dL, AST/ALT < 2.5 x ULN

Exclusion Criteria:

* Patient with progressive disease during first line chemotherapy with a platinum/taxane combination will be excluded.
* Patients must not have clinically significant autoimmune disease that requires treatment with immunosuppressant medications.
* Because of compromised cellular immunity and limited capacity to respond to vaccination, patients who are HIV+ will be excluded.
* Patients must not have serious intercurrent illness such as infection requiring IV antibiotics, or significant cardiac disease characterized by significant arrhythmia, unstable ischemic coronary disease or congestive heart failure.
* Pregnant and/or lactating women will be excluded. Premenopausal patients will undergo pregnancy testing when indicated. Women will practice effective birth control while receiving protocol treatment.
* Patients with a history of clinically significant venous thromboembolism will be excluded.
* Active second malignancy, aside from basal cell or squamous cell carcinoma of the skin (i.e. malignancy not treated with curative intent or diagnosis within the past 2 years)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2008-08; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To determine if cellular immunity is induced by serial vaccination with DC/tumor fusion cells, when given with GM-CSF alone, or the combination of GM-CSF and imiquimod in this patient population. | 2 years

SECONDARY OUTCOMES:
To assess toxicity associated with vaccination with DC/tumor fusion when given with GM-CSF and imiquimod. | 2 years
To assess clinical response to vaccination with DC/tumor fusion when given with GM-CSF and imiquimod. | 2 years
To correlate immunologic response following vaccination with measures of patient cellular immune function and phenotypic characteristics of the vaccine preparation. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David Avigan, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts